CLINICAL TRIAL: NCT02322593
Title: An Open-label Randomized Multi-center Phase III Study of TAS-118 Plus Oxaliplatin Versus S-1 Plus Cisplatin as First-line Therapy in Patients With Advanced Gastric Cancer
Brief Title: Phase III Study of TAS-118 Plus Oxaliplatin Versus S-1 Plus Cisplatin in Patients With Advanced Gastric Cancer
Acronym: SOLAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Collaborators: Yakult Honsha Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10056040
Record Dates: First submitted 2014-12-12; First posted 2014-12-23 (Estimated); Results first posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-11

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Gastrointestinal Diseases; Gastrointestinal Neoplasms; First Line Treatment; Antineoplastic Agents
MeSH Terms: conditions — Stomach Neoplasms; Gastrointestinal Diseases; Gastrointestinal Neoplasms | interventions — Oxaliplatin; S-1 plus cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAS-118/Oxaliplatin (Experimental): TAS-118 plus Oxaliplatin
  Interventions: Drug: TAS-118 plus Oxaliplatin
- S-1/Cisplatin (Active Comparator): S-1 plus Cisplatin
  Interventions: Drug: S-1 plus Cisplatin

INTERVENTIONS:
Drug: TAS-118 plus Oxaliplatin
  Arms: TAS-118/Oxaliplatin
Drug: S-1 plus Cisplatin
  Arms: S-1/Cisplatin

SUMMARY:
The purpose of this trial is to evaluate the efficacy of TAS-118 plus Oxaliplatin compared with S-1 plus Cisplatin in overall survival in patients with advanced gastric cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients who are diagnosed as gastric cancer.
* No prior treatment for gastric cancer.
* Negative or unknown for HER2 testing.
* ECOG performance status of 0 or 1.

Key Exclusion Criteria:

* Unmanageable diarrhea.
* Current peripheral sensory neuropathy or paresthesia.
* Pregnant or lactating female.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (3):
  - Taiho Pharmaceutical Co., Ltd selected site, Ibaraki
  - Taiho Pharmaceutical Co., Ltd selected site, Kumamoto
  - Taiho Pharmaceutical Co., Ltd selected site, Tokyo
- Taiho Pharmaceutical Co., Ltd selected site, Seoul, South Korea

REFERENCES:
- [Derived] Kang YK, Chin K, Chung HC, Kadowaki S, Oh SC, Nakayama N, Lee KW, Hara H, Chung IJ, Tsuda M, Park SH, Hosaka H, Hironaka S, Miyata Y, Ryu MH, Baba H, Hyodo I, Bang YJ, Boku N. S-1 plus leucovorin and oxaliplatin versus S-1 plus cisplatin as first-line therapy in patients with advanced gastric cancer (SOLAR): a randomised, open-label, phase 3 trial. Lancet Oncol. 2020 Aug;21(8):1045-1056. doi: 10.1016/S1470-2045(20)30315-6. Epub 2020 Jul 16. PMID 32682457

RESULTS

PARTICIPANT FLOW:
Groups:
- TAS-118/Oxaliplatin: TAS-118 plus Oxaliplatin
  L-OHP was administered intravenously at dose of 85 mg/m2 on day 1, and TAS-118 were administered 30-60 mg orally twice daily for 7 days (day 1 through day 7), repeated every 2 weeks. Treatment was continued during the study period unless any of Study Treatment Discontinuation Criteria was met.
- S-1/Cisplatin: S-1 plus Cisplatin
  CDDP was administered intravenously at dose of 60 mg/m2 on day 1 (Korea) or day 8 (Japan), and S-1 were administered 40-60 mg orally twice daily for 21 days (day 1 through day 21), repeated every 5 weeks (rest period can be shorten from 14 days to 7 days). Treatment was continued during the study period unless any of Study Treatment Discontinuation Criteria was met.
Period: Overall Study
Arm/Group | TAS-118/Oxaliplatin | S-1/Cisplatin
Started | 356 | 355
Completed | 356 | 355
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS)：Patients in AT population who have advanced gastric cancer at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAS-118/Oxaliplatin | S-1/Cisplatin | Total
Number analyzed (Participants) | 347 | 334 | 681
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 201 | 194 | 395
  >=65 years | 146 | 140 | 286
Age, Continuous [Median (Full Range); unit: years] | 62.0 [21 to 79] | 62.0 [26 to 80] | 62.0 [21 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 116 | 212
  Male | 251 | 218 | 469
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 347 | 334 | 681
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 347 | 334 | 681
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 221 | 212 | 433
  South Korea | 126 | 122 | 248

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The primary endpoint was OS, which was defined as the time from the date of randomization to the date of death from any cause. Surviving patients were censored at the cutoff date or last contact date if lost to follow-up, or upon withdrawal of consent.
Time Frame: A survival follow-up was required every 12 weeks from the date of randomization to the date of death from any cause, whichever came first, assessed up to 38 months.
Population: Full Analysis Set (FAS)：Patients in AT population who have advanced gastric cancer at randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TAS-118/Oxaliplatin | S-1/Cisplatin
Number analyzed (Participants) | 347 | 334
Months | 16.0 [13.8 to 18.3] | 15.1 [13.6 to 16.4]
Statistical Analysis 1: Comparison: TAS-118/Oxaliplatin; Test type: Superiority; p = 0.039, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.69 to 0.99], Standard Error of Mean 0.091

2. Secondary Outcome: Progression-free Survival
Description: PFS was defined as the time from the date of randomization to the date of disease progression (assessed by each investigator) or death from any cause, whichever came first.
Time Frame: A radiographic imaging examination using CT or MRI was repeated every 6 weeks. Tumor assessments were performed from the date of randomization to the date of disease progression or death from any cause, whichever came first.
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TAS-118/Oxaliplatin | S-1/Cisplatin
Number analyzed (Participants) | 347 | 334
Months | 7.1 [6.8 to 8.3] | 6.4 [5.6 to 6.9]
Statistical Analysis 1: Comparison: TAS-118/Oxaliplatin; Test type: Superiority; p = 0.0045, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.66 to 0.93], Standard Error of Mean 0.086

3. Secondary Outcome: Time to Treatment Failure
Description: TTF was defined as the time from the date of randomization to the date of the last administration of the study drug. Patients on study treatment were censored at the date of the last administration or the cutoff date, whichever came earlier.
Time Frame: From the date of randomization to the date of the last administration of the study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TAS-118/Oxaliplatin | S-1/Cisplatin
Number analyzed (Participants) | 347 | 334
Months | 6.1 [5.6 to 6.7] | 5.3 [4.7 to 6.2]
Statistical Analysis 1: Comparison: TAS-118/Oxaliplatin; Test type: Superiority; p = 0.011, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.70 to 0.96], Standard Error of Mean 0.078

4. Secondary Outcome: Overall Response Rate
Description: ORR was defined as the proportion of patients with the best unconfirmed overall response of complete response (CR) or partial response (PR) in patients with measurable lesions
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 42 months.
Population: Tumor Response (TR) Evaluable Population： Patients in FAS population presenting measurable lesions (at least one target lesion), evaluated for tumor responses at least once during treatment with the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-118/Oxaliplatin | S-1/Cisplatin
Number analyzed (Participants) | 211 | 212
Participants | 155 | 106
Statistical Analysis 1: Comparison: TAS-118/Oxaliplatin; Test type: Superiority; p < 0.001, Fisher Exact

5. Secondary Outcome: Disease Control Rate
Description: DCR was defined as the proportion of patients with CR, PR, or stable disease in patients with measurable lesions.
Time Frame: as for outcome 4
Population: TR Evaluable Population：
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-118/Oxaliplatin | S-1/Cisplatin
Number analyzed (Participants) | 211 | 212
Participants | 197 | 187
Statistical Analysis 1: Comparison: TAS-118/Oxaliplatin; Test type: Superiority; p = 0.092, Fisher Exact

ADVERSE EVENTS:
Time Frame: From the time a patient signed informed consent until 30 day safety follow-up visit or initiation of new anticancer treatment, whichever was earlier, an average assessed up to 42 months.
Description: An adverse event (AE) is any untoward medical condition that occurs in a patient while participating in a clinical study and does not necessarily have a causal relationship with the use of the product. Treatment emergent adverse events are AEs that occur from the initiation of any study medication administration, and do not necessarily have a causal relationship to the use of the study medication.
Arm/Group | TAS-118/Oxaliplatin | S-1/Cisplatin
All-Cause Mortality (participants affected / at risk) | 22/352 | 8/348
Serious Adverse Events (participants affected / at risk) | 155/352 | 159/348
Other Adverse Events (participants affected / at risk) | 344/352 | 328/348
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAS-118/Oxaliplatin (N=352) | S-1/Cisplatin (N=348)
Anaemia (Blood and lymphatic system disorders) | 2 | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 6
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 1
Rhegmatogenous retinal detachment (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 10 | 9
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 5 | 8
Cheilitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 14 | 8
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 5 | 2
Enterocolitis (Gastrointestinal disorders) | 3 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 3 | 2
Gastric perforation (Gastrointestinal disorders) | 0 | 3
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 7 | 5
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 11 | 6
Obstruction gastric (Gastrointestinal disorders) | 3 | 8
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal stenosis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 4 | 1
Oesophageal discomfort (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric stenosis (Gastrointestinal disorders) | 2 | 4
Large intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Rectal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 4 | 2
Condition aggravated (General disorders) | 1 | 0
Death (General disorders) | 1 | 1
Fatigue (General disorders) | 3 | 4
Malaise (General disorders) | 2 | 2
Mucosal inflammation (General disorders) | 1 | 1
Mucous membrane disorder (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 10 | 5
Disease progression (General disorders) | 5 | 1
Complication associated with device (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2
Jaundice (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 3 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Dacryocystitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 8 | 7
Pneumonia herpes viral (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urethritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 1
Cytomegalovirus enterocolitis (Infections and infestations) | 1 | 0
Cytomegalovirus enteritis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Enteritis infectious (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 3
Biliary tract infection (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Fractured ischium (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 6
Platelet count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 6
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 39 | 32
Hypophagia (Metabolism and nutrition disorders) | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 2
Dementia (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Presyncope (Nervous system disorders) | 0 | 2
Seizure (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Embolic cerebral infarction (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 4 | 8
Renal disorder (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2
Renal impairment (Renal and urinary disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Adnexal torsion (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 2
Infarction (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAS-118/Oxaliplatin (N=352) | S-1/Cisplatin (N=348)
Anaemia (Blood and lymphatic system disorders) | 94 | 96
Leukopenia (Blood and lymphatic system disorders) | 14 | 19
Neutropenia (Blood and lymphatic system disorders) | 50 | 53
Lacrimation increased (Eye disorders) | 41 | 37
Abdominal pain (Gastrointestinal disorders) | 46 | 30
Constipation (Gastrointestinal disorders) | 80 | 90
Diarrhoea (Gastrointestinal disorders) | 189 | 134
Dyspepsia (Gastrointestinal disorders) | 20 | 13
Nausea (Gastrointestinal disorders) | 200 | 186
Stomatitis (Gastrointestinal disorders) | 148 | 88
Vomiting (Gastrointestinal disorders) | 100 | 70
Fatigue (General disorders) | 116 | 106
Malaise (General disorders) | 77 | 76
Oedema (General disorders) | 9 | 26
Oedema peripheral (General disorders) | 21 | 27
Pyrexia (General disorders) | 45 | 32
Alanine aminotransferase increased (Investigations) | 45 | 20
Aspartate aminotransferase increased (Investigations) | 50 | 19
Blood creatinine increased (Investigations) | 6 | 33
Neutrophil count decreased (Investigations) | 90 | 115
Platelet count decreased (Investigations) | 103 | 76
Weight decreased (Investigations) | 78 | 41
White blood cell count decreased (Investigations) | 45 | 76
Blood alkaline phosphatase increased (Investigations) | 27 | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 40 | 25
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 14
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 19
Decreased appetite (Metabolism and nutrition disorders) | 234 | 216
Dizziness (Nervous system disorders) | 18 | 34
Dysgeusia (Nervous system disorders) | 112 | 82
Neuropathy peripheral (Nervous system disorders) | 21 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 242 | 54
Hiccups (Respiratory, thoracic and mediastinal disorders) | 19 | 62
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 23
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 60 | 27
Rash (Skin and subcutaneous tissue disorders) | 18 | 19
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 63 | 50
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 32 | 17
Vascular pain (Vascular disorders) | 32 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT02322593/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT02322593/SAP_001.pdf